CLINICAL TRIAL: NCT06715215
Title: Role of Acute Phase Proteins In Diagnosis of Immune Thrombocytopenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rana Mohamed Abdelhameed, Resident of clinical pathology department, Sohag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-11-13MS
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- age and sex matched thrombocytopenic patients other than ITP. (Active Comparator): Causes of decreased platelets count other than immune thrombocytopenia
  Interventions: Diagnostic Test: Acute phase proteins
- acute ITP patients (Active Comparator): Patients diagnosed as acute thrombocytopenia
  Interventions: Diagnostic Test: Acute phase proteins
- chronic ITP patients . (Active Comparator): Patients diagnosed as chronic thrombocytopenia
  Interventions: Diagnostic Test: Acute phase proteins

INTERVENTIONS:
Diagnostic Test: Acute phase proteins — Assessment of acute phase proteins levels in patients diagnosed with immune thrombocytopenia

SUMMARY:
Immune thrombocytopenia (ITP) are antibody-mediated disorders in which platelets are destroyed mainly through activating immunoglobulin (IgG) Fc receptors on phagocytes in the spleen and liver, eventually resulting in thrombocytopenia Acute phase proteins (APP) are inflammation markers that exhibit significant changes in serum concentration during inflammation. These are also important mediators produced in the liver during acute and chronic inflammatory states. Acute phase reactants can be classified as positive or negative, depending on their serum concentrations during inflammation. Positive acute phase reactants are upregulated, and their concentrations increase during inflammation. Negative acute phase reactants are downregulated, and their concentrations decrease during inflammation. Positive acute phase proteins include procalcitonin, C-reactive protein, ferritin, fibrinogen, hepcidin, and serum amyloid A. Negative acute phase reactants include albumin, prealbumin, transferrin, retinol-binding protein, and antithrombin CRP is now well established as a major acute phase protein and is used in daily clinical practice as a sensitive biomarker for infection and inflammation, with its level increasing from <0.05 to >500 mg/L after acute infections. CRP is produced by hepatocytes, in response to inflammatory cytokines such as interleukin (IL)-6 and IL-1, with serum concentrations rising to >5 mg/L after 6 hours and peaking after ∼48 hours. In healthy young adult volunteer blood donors, the median concentration of CRP was found to be ∼0.8 mg/L CRP levels are useful as a clinical diagnostic tool for infection, and it is a common knowledge that ITP is triggered by viral infection that precedes the clinical picture of ITP by a few days to a few weeks Procalcitonin (PCT) is used as a reliable inflammatory biomarker with high sensitivity and specificity ferritin was confirmed as an inflammation and infection biomarker in the diagnosis of viral and bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with platelet less than 100 × 109/L diagnosed as immune thrombocytopenia by bone marrow findings .

Age of patients : from 1 year to 50 years.

Exclusion Criteria:

* - Other causes of thrombocytopenia as:

  * Hypersplenism.
  * Bone marrow diseases including : aplastic anemia, leukemia and myelodysplastic syndromes.
  * Cancer treatments like chemotherapy and radiation therapy.
  * Exposure to toxic chemicals as arsenic and benzene.
  * Medications to treat bacterial infections (antibiotics)and treat seizures or blood thinner heparin.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute phase proteins | 2 years
  By taking serum samples from pateints and measure acute phase proteins levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Sahag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gruys E, Toussaint MJ, Niewold TA, Koopmans SJ. Acute phase reaction and acute phase proteins. J Zhejiang Univ Sci B. 2005 Nov;6(11):1045-56. doi: 10.1631/jzus.2005.B1045. PMID 16252337
- [Background] Zeller B, Rajantie J, Hedlund-Treutiger I, Tedgard U, Wesenberg F, Jonsson OG, Henter JI; NOPHO ITP. Childhood idiopathic thrombocytopenic purpura in the Nordic countries: epidemiology and predictors of chronic disease. Acta Paediatr. 2005 Feb;94(2):178-84. doi: 10.1111/j.1651-2227.2005.tb01887.x. PMID 15981751
- [Background] Semple JW, Italiano JE Jr, Freedman J. Platelets and the immune continuum. Nat Rev Immunol. 2011 Apr;11(4):264-74. doi: 10.1038/nri2956. PMID 21436837
- [Background] Sullivan PS, Hanson DL, Chu SY, Jones JL, Ciesielski CA. Surveillance for thrombocytopenia in persons infected with HIV: results from the multistate Adult and Adolescent Spectrum of Disease Project. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Apr 1;14(4):374-9. doi: 10.1097/00042560-199704010-00011. PMID 9111481